CLINICAL TRIAL: NCT01940055
Title: A Phase II, Pilot-Randomized Clinical Trial to Study the Effect of a Novel Dual-Task Exercise Program for Balance, Mobility and Cognition in Community Dwelling Older Adults
Brief Title: The Effect of a Novel Dual-Task Exercise Program for Balance, Mobility and Cognition in Community Dwelling Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Not yet recruiting
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2013-12

CONDITIONS: Aging
Keywords: Balance; Gait; Instrumented Treadmill; Recumbent cycle; Cognitive games

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Dual Task Treadmill Walking Exercise Program
  Interventions: Behavioral: Dual task treadmill walking exercise program
- Control group (Active Comparator): Dual task recumbent cycling exercise program
  Interventions: Behavioral: Dual task recumbent cycling exercise program

INTERVENTIONS:
Behavioral: Dual task treadmill walking exercise program — Participants will receive 5 minute warm up and cool down session followed by a 30 minute dual task program which includes treadmill walking while playing brain fitness or cognitive games. Rest periods will be provides to the participants. Treadmill speed will be set so as to not exceed 60% of maximum heart rate. Heart rate and perceived excretion( per the Borg 1-10) will be measured at 5 minutes of interval.
  Arms: Experimental group
Behavioral: Dual task recumbent cycling exercise program — Participants will receive a 5 minute warm up and cool down session followed by a 30 minute dual task exercise program which includes recumbent cycling while playing brain fitness or cognitive games. Rest periods will be provides to the participants. Recumbent cycling speed will be set so as to achieve 60% of maximum heart rate. Heart rate and perceived excretion( per the Borg 1-10) will be measured at 5 minutes of interval.
  Arms: Control group

SUMMARY:
Goal:

The development of a Treadmill Rehabilitation Platform (TRP) for task-orientated rehabilitation that provides an adapted, blended approach among older adults with balance, mobility, and cognitive impairments.

Study Objective:

Examine the feasibility and benefits of a novel dual-task intervention to address mobility and cognitive decline with age using engaging interactive video games during treadmill walking and recumbent cycling.This will include evaluation of the effects of two interventions, one using treadmill walking and the second a recumbent cycle ergometer on

1. Core balance
2. Cardiac fitness, exercise endurance
3. Gaze control
4. Gait performance measure (walking stability and spatial-temporal gait parameters)
5. Specific executive cognitive function (processing speed, cognitive inhibition, working memory)
6. Dual task function during treadmill walking

Hypothesis:

1. Dual-task exercise program will improve core balance and walking function to a greater extent in the Treadmill walking group compared to recumbent cycle group.
2. Executive function will improve equally in both the treadmill walking and recumbent cycle group.
3. Dual task exercise programs will have significant effect on gaze stability and cardiac fitness equally for both the treadmill and recumbent cycling groups.

DETAILED DESCRIPTION:
Study design: A phase II, Pilot-Randomized clinical trial. Sample size will be 15 volunteer older adults for each group, aged between 70-80 years old living in the community and attending the Reh-Fit center for exercise.

Method:

Recruitment:

Individuals attending the Reh-Fit center for exercise and physical activity. This will be coordinated and organized by staff at Reh-Fit center who will inform their members about this research study.

Interventions:

Each participant will receive a 45 minute program of combined exercise and cognitive activities twice a week for 10 weeks.

One group will receive the dual-task treadmill walking program (DT-TW) and the 2nd group will receive the dual-task recumbent cycling program (DT-RC). Both programs will contain the same cognitive activities delivered through interactive "cognitive" video games.

Dual-task treadmill walking program (DT-TW):

* 5 minute warm up and cool down at a speed equivalent to a comfortable walking speed.
* 30 minutes of dual-task treadmill walking at 2-3 speed levels . Speed will be selected NOT to exceed 60% of Max-HR, Heart rate (HR), blood. Heart rate, blood pressure and Perceived exertion (Per the Borg 1-10 scale) will be measured at 5 minute intervals.

Dual-task recumbent cycling program (DT-RC)

* 5 minute warm up and cool down at a per-determined speed and resistance where heart rate wold not exceed 40 percent of age maximum ( 220 minus age)
* 30 minutes of dual-task (treadmill walking group or recumbent cycle group) training, while performing concurrent cognitive games with a few minutes of rest periods in between as required. The intensity of cycling will be selected achieve 50- 60% of Max-HR. Heart rate, blood pressure and Perceived exertion (Per the Borg 1-10 scale) will be measured at 5 minute intervals

For each participant five to eight computer games will be selected to play during walking or cycling from a collection of over 60 purchased form Big Fish Games (www.bigfishgames.com).

A commercial motion mouse (Gyration Air Mouse, USA) was secured to a head band and used as the computer input device to control on-screen cursor motion with head rotation (left-right). This motion Mouse has inertial sensors used to derive angular position signals. With this simple method, seamless and responsive hands-free interaction with most computer applications is made possible.

The computer games involve goal- directed cognitive activities which includes a mix of (a) precision movements to interact with game targets, (b) the presence of distractors, (c) search and matching tasks, and (d) working memory.

Data Analysis and Outcome Measures:

Demographic and clinical data: Age, sex, fall history, Mini Mental score Examination (MMSE) greater than 24.

The Community Health Activities Model Program for Seniors questionnaire (CHAMPS).

Primary outcomes:

Cardiac fitness measured by Young Men's Christian Association (YMCA) Cycle Ergometer Sub-maximal test (ACSM's Guidelines for Exercise Testing and . During the test, heart rate (HR), blood pressure (BP), revolution per minute (RPM) and rate of perceived exertion (RPE) were recorded at 5 minutes interval (Borg, 1982).

Validated performance-based measures of balance; (i) Clinical Test of Sensory Integration of Balance , (ii) Five-Time Sit-to-Stand Test.

Walking endurance will be measured using the 6-minute walk test.

Spatial and Temporal Gait Variables will be measured during treadmill walking at a fixed speed of 0.9 meter per second. A treadmill instrumented with a Force Sensory Array(FSA) pressure mat (Vista Medical, Ca) will be used for this purpose . Each participant will walk for two minutes and the following variables (average and coefficient of variation of 60 consecutive steps); will be determined: stance duration, swing time, step time, step length and step width.

Dual task walking performance: A custom computer application which works with the Gyration motion mouse was developed for this purpose. The cognitive game task was similar to the Useful Field of View test the (UFOV). The goal of the test game is to move a paddle (game sprite) to catch falling bright circle objects (targets) moving vertically top to bottom, and to avoid other shape (or colors) game objects (dis-tractors). The objects appear at user defined fixed intervals (e.g. 2 seconds) and at random locations on the monitor. The game is instrumented with an assessment module. This generates a logged game file recording (80 Hz) the following signals associated with player performance with respect to game events: (i) time index and coordinates of each game object and (ii) position coordinates of the game paddle (slaved to head rotation). Features of the test game events provide a basis for objective quantification of cognitive functions, which include. (i) game success rate (percentage of target caught), (ii) average motor response time (time from appearance of the target to start of the paddle movement), (iii) average movement execution time (iv) movement efficiency. The cognitive game task is first performed in standing (single tasks) and then during treadmill waking at 0.9 m/s (dual-task walking condition). The difference in spatial -temporal gait variables during walk alone ( as describe above) and dual task walking condition will be used to index dual-task performance.

Gaze Stability Test: A custom computer application was developed for this purpose. This consists of tracking a bright visual target moving horizontally left and right on a computer display at fixed amplitude (80% of the monitor width) at a frequency of 0.4 Hz. A 70 m monitor was used, positioned at eye-level, 100 cm away from the participant. This results in head horizontal rotations of between 30 to 40 degrees, left and right of center. The test procedure involves a closed loop tracking task (with respect to head). In this task two cursors of different colors appear on the monitor. One is the target cursor and the 2nd cursor is slaved to head rotation via the head mounted motion mouse. The task goal is to overlap the two cursors during the cyclic left-to-right cursor motion. In this task foveation is necessary to determine the amount of overlap (error) between the target cursor and the head cursor.

Nero-psychological tests: We will use the Standardized Nero-psychological tests targeting executive functions: This includes a test battery of three executive functions (Trial Making Test A-B, verbal fluency, and visual Search.). Also, The National Institutes of Health (NIH) toolbox cognitive tests, targeting executive functions that include dimensional change card sort.

1. Trial Making test (A & B): It is a valid and reliable well-established test, which is a valid measure to target speed of processing, response inhibition and task-switching. This test is graded by time. It has been used widely in clinical evaluations for the assessment of deficits in cognitive function. It is administered in two parts: 1) Trial Making test form A, the subject is required to draw lines sequentially connecting numbered circles arranged randomly on a page as quickly as possible; 2) Trial Making test form B is a more demanding task as it requires the subject to connect circles containing numbers and letters in an alternating sequence.
2. Verbal fluency: It is a test of working memory and language in which participants have to say as many words as possible from a category in a given time (usually 60 seconds). The test includes both semantic and phonemic sections, and has been shown to be highly reliable and valid among elderly population.
3. Visual search test: It is a test of speed of processing, cognition inhibition and attention in which the participants have to look for a target stimulus among dis-tractor stimuli (usually 60 seconds). The test measures both reaction time and the number of selected items. It has been shown to be reliable and valid measure among elderly.
4. Dimensional change card sort: It is a test of working memory and cognitive inhibition in which the participants are asked to match sets of two test pictures that differ in color to target pictures (usually 10 seconds). The test measures both reaction time and the number of selected items.

Participants will be assessed by a blinded assessor prior to beginning the intervention and within one week of completing the 10 week program. Pre and post intervention assessment will be spread over two days, each lasting approximately 60 minutes with ample rest periods. Performing the balance and treadmill walking assessments while performing concurrent cognitive tasks may be difficult and participants may lose their balance. The treadmill is equipped with safety side rails which are within easy reach, and participants will be fitted with a safety harness secured above to a support system. Also during all tests, a Physical Therapist will stand behind or beside the participants to provide assistance if required.

Statistical Analysis:

We will compare and test the difference in baseline values of demographic data, walking ability and the validated performance-based measures of balance between groups circuits training with Mann-Whitney U test for ordinal scale outcomes and student's t-test for independent groups assuming equal variances.

A mixed model repeated measure (ANOVA) will be used to examine the within group and between group effects on the dependent variables representing cardiac fitness, core balance, walking stability and dual-task walking performance, , gaze stability, and executive cognitive function parameters (Hypothesis 1); Executive function (Hypothesis 2); Gaze control and cardiac fitness (Hypothesis 3).

ELIGIBILITY:
Inclusion criteria:

1. Age between 70-80 years old.
2. Independent community dwelling
3. Walk 400 meters without a walking aid or using a single-point stick only.
4. Mini mental status test score greater than 24
5. Experiencing no more than one fall in the previous 12 months.
6. Having concerns about their balance which is based on participants' positive response to the question: "Are you concerned about your balance?"
7. Adequate hearing and vision

Exclusion Criteria:

1. Clinical diagnosis of dementia and a Mini Mental State Exam score less than 24,
2. Self-reported diagnosis or history of (i) stroke, traumatic brain injury or other neurological disorders such as Parkinson's disease and Vestibular disorders, (ii) cardiac disease, and (iii) muscular-skeletal injuries or orthopaedic diseases such as acute lower back or lower extremity pain, peripheral neuropathy, advanced hip/knee osteoporosis.
3. Any recent medical illness that would affect their balance or ability to walk for a period of at least 6 minutes.

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Dual task function during walking | Pre and post intervention of 10 weeks
  Walking on at treadmill at a speed of 0.9 m/s while performing a cognitive game task simultaneously i.e the participants move a paddle (game sprite to catch bright circle objects(targets)moving vertically top to bottom, avoiding other shape(or colors) game objects (dis-tractors). This test game provides an objective quantification of cognitive functions like (i) Game success rate (percentage of target caught), (ii) average motor response time (time from appearance of the target to start of the paddle movement), (iii) average movement execution time (iv) movement efficiency .
Executive function | Pre and post intervention of 10 weeks
  Neuropsychological tests:Trail making test (A and B), Verbal Fluency, Visual Search and the dimensional change card sort test
Core Balance | Pre and post intervention of 10 weeks
  I t will be measured by performing a) Clinical Test of Sensory Integration of Balance and b) Five - Time Sit-to-Stand Test
Spatial - temporal gait variables | Pre and post intervention of 10 weeks
  It will be measured by asking the participants to walk on a treadmill for 2 minutes which is instrumented with a pressure mat at a speed of 0.9 m/s. Average and coefficient of variation will be obtained for the following parameters: swing time, step time, step length and step width.
Cardiac fitness | Pre and post Intervention of 10 weeks
  Cycle ergometer Submaximal Test will be performed measuring the heart rate, blood pressure, revolution per minute and rate of perceived exertion at an interval of 5 minutes.

SECONDARY OUTCOMES:
6- Minute walk test | Pre and post intervention of 10 weks
CHAMPS Questionnaire | Post intervention of 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Akshata V Nayak, MSc Student, Principal Investigator — University of Manitoba; Rehab Alhasani, MSc Student, Principal Investigator — University of Manitoba; Tony Szturm, PT,PhD, Principal Investigator — University of Manitoba; Geri Brousseau, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Reh Fit Center, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Szturm T, Betker AL, Moussavi Z, Desai A, Goodman V. Effects of an interactive computer game exercise regimen on balance impairment in frail community-dwelling older adults: a randomized controlled trial. Phys Ther. 2011 Oct;91(10):1449-62. doi: 10.2522/ptj.20090205. Epub 2011 Jul 28. PMID 21799138
- [Background] Lockery D, Peters JF, Ramanna S, Shay BL, Szturm T. Store-and-feedforward adaptive gaming system for hand-finger motion tracking in telerehabilitation. IEEE Trans Inf Technol Biomed. 2011 May;15(3):467-73. doi: 10.1109/TITB.2011.2125976. PMID 21536526
- [Background] Szturm T, Maharjan P, Marotta JJ, Shay B, Shrestha S, Sakhalkar V. The interacting effect of cognitive and motor task demands on performance of gait, balance and cognition in young adults. Gait Posture. 2013 Sep;38(4):596-602. doi: 10.1016/j.gaitpost.2013.02.004. Epub 2013 Mar 9. PMID 23477841